CLINICAL TRIAL: NCT01529047
Title: RTC of Web Versus In-Person SUD and Comorbidity Treatment
Brief Title: Web-based vs In-person Personalized Feedback Intervention for Comorbid Substance Use and Disordered Gambling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mary Larimer, Professor, Psychiatry & Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35898; R01DA025051 (NIH)
Record Dates: First submitted 2012-02-03; First posted 2012-02-08 (Estimated); Last update posted 2023-06-27 (Actual); Status verified 2016-06

CONDITIONS: Gambling; Alcohol Consumption; Cannabis
MeSH Terms: conditions — Gambling; Alcohol Drinking; Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- In-person PFI (Experimental): In-person personalized feedback intervention
  Interventions: Behavioral: Personalized Feedback Intervention
- Web-based PFI (Experimental): Web-based personalized feedback intervention
  Interventions: Behavioral: Personalized Feedback Intervention
- Assessment Only (No Intervention): Complete online survey assessments only.

INTERVENTIONS:
Behavioral: Personalized Feedback Intervention — Printed or electronic form containing personalized information about health-relevant behaviors
  Arms: In-person PFI; Web-based PFI

SUMMARY:
Rates of gambling and substance use behaviors are elevated among emerging adults (ages 18-24), and these behaviors are individually and jointly associated with a host of negative consequences. Evidence suggests there is significant overlap between these behaviors as well as comorbidity of associated mental disorders (i.e., pathological gambling and substance abuse/dependence). Prior research suggests that a brief in-person delivered personalized feedback intervention (PFI) may be an effective method of reducing these behaviors and their associated consequences among emerging adults. Thus, the purpose of this study is to determine the relative efficacy of an in-person delivered PFI versus a Web-based PFI in reducing gambling, alcohol and marijuana use behaviors and related-consequences in a sample of emerging adults, as well as explore potential moderators and mediators of intervention efficacy and the longevity of intervention effects (over a period of 18-months).

ELIGIBILITY:
Inclusion Criteria:

* Endorse disordered gambling behavior (including 1 or more consequence)
* Meet diagnostic criteria for one or more substance use disorder

Exclusion Criteria:

* Not meeting inclusion criteria

Ages: 17 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 361 (Actual)
Dates: Start 2010-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
gambling behavior and consequences | across 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Larimer, Ph.D., Principal Investigator — University of Washington Dept of Psychiatry & Behavioral Sciences
Locations (1):
- University of Washington, Seattle, Washington, United States